CLINICAL TRIAL: NCT01989910
Title: An Open Label, Randomized, Parallel Design Estimation Pilot Study to Compare the Efficacy and Safety of Raltegravir-based Versus Efavirenz-based Combination Therapy in Treatment-naïve Patients With HIV-1 Infection
Brief Title: Compare the Efficacy and Safety of Raltegravir Versus Efavirenz Combination Therapy in Treatment-naïve HIV-1 Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSD-MISP-39299; TVGH-IRB-2013-07-030B (Other: TaipeiVGH)
Record Dates: First submitted 2013-10-22; First posted 2013-11-21 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-10

CONDITIONS: HIV-1 Infection
Keywords: Efavirenz; Raltegravir; Combination antiretroviral therapy
MeSH Terms: interventions — Raltegravir Potassium; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Raltegravir (Active Comparator): Raltegravir 400mg oral twice daily
  Interventions: Drug: Efavirenz
- Efavirenz (Active Comparator): Efavirenz 600mg oral at bedtime
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 400mg oral twice daily
  Other Names: Isentress
  Arms: Efavirenz
Drug: Efavirenz — Efavirenz 600mg oral at bedtime
  Other Names: Stocrit
  Arms: Raltegravir

SUMMARY:
A pilot study to compare the efficacy and safety of raltegravir-based versus efavirenz-based combination therapy in treatment-naïve patients with HIV-1 infection.

DETAILED DESCRIPTION:
A single-center, prospective, randomized, open label, parallel study to compare the efficacy and safety of raltegravir-based versus efavirenz-based plus optimal nucleoside reverse-transcriptase inhibitors(NRTIs) backbone combination therapy in treatment-naïve patients with HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are infected with HIV-1
* Patients have not yet received any treatment for HIV
* Patients with HIV viral RNA exceeds 5000 copies per ml
* Ages at least 20 years

Exclusion Criteria:

* Patients with acute or decompensated chronic hepatitis
* Patients with chronic hepatitis and serum aminotransferase concentrations are more than five times the upper limit of the normal range
* Patients with renal insufficiency (need dialysis or have serum creatinine concentrations of more than twice the upper limit of the normal range
* Patients with any medical disorder that the use of study medications is contraindicated
* Pregnant or breastfeeding women
* Patients who are lack of expectation to maintain assigned study medication during study period
* Patients who have received therapy with investigational drugs in the previous 3 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wing Wai Wong, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Division of Infectious Diseases, Taipei Veterans General Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Lennox JL, DeJesus E, Lazzarin A, Pollard RB, Madruga JV, Berger DS, Zhao J, Xu X, Williams-Diaz A, Rodgers AJ, Barnard RJ, Miller MD, DiNubile MJ, Nguyen BY, Leavitt R, Sklar P; STARTMRK investigators. Safety and efficacy of raltegravir-based versus efavirenz-based combination therapy in treatment-naive patients with HIV-1 infection: a multicentre, double-blind randomised controlled trial. Lancet. 2009 Sep 5;374(9692):796-806. doi: 10.1016/S0140-6736(09)60918-1. Epub 2009 Aug 3. PMID 19647866
- [Background] Steigbigel RT, Cooper DA, Teppler H, Eron JJ, Gatell JM, Kumar PN, Rockstroh JK, Schechter M, Katlama C, Markowitz M, Yeni P, Loutfy MR, Lazzarin A, Lennox JL, Clotet B, Zhao J, Wan H, Rhodes RR, Strohmaier KM, Barnard RJ, Isaacs RD, Nguyen BY; BENCHMRK Study Teamsa. Long-term efficacy and safety of Raltegravir combined with optimized background therapy in treatment-experienced patients with drug-resistant HIV infection: week 96 results of the BENCHMRK 1 and 2 Phase III trials. Clin Infect Dis. 2010 Feb 15;50(4):605-12. doi: 10.1086/650002. PMID 20085491
- [Background] Young B, Vanig T, Dejesus E, Hawkins T, St Clair M, Yau L, Ha B, Shield Study Team. A pilot study of abacavir/lamivudine and raltegravir in antiretroviral-naive HIV-1-infected patients: 48-week results of the SHIELD trial. HIV Clin Trials. 2010 Sep-Oct;11(5):260-9. doi: 10.1310/hct1105-260. PMID 21126956

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raltegravir | Efavirenz
Started | 53 | 54
Completed | 51 | 54
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Efavirenz | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [27 to 40] | 33 [31 to 43] | 32 [29 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 50 | 52 | 102
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 51 | 54 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline VL >100,000 copies/mL [Count of Participants; unit: Participants] | 27 | 28 | 55

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Patients Who Can Achieve of Less Than 20 HIV RNA Copies Per ml at Week 48 of Both Arms.
Description: Virological response to achieve HIV RNA copies <20 copies/mL at week 48 of both arms.
Time Frame: At week 48 of both arms
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 51 | 54
Participants | 41 | 36

2. Secondary Outcome: The Proportion of Patients With Achievement of Less Than 400 HIV RNA Copies Per ml at Week 48 for Both Arms.
Description: Virological response to achieve HIV RNA copies <400 copies/mL at week 48 of both arms.
Time Frame: At week 48 of both arms
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 51 | 54
Participants | 41 | 36

3. Secondary Outcome: The Change From Baseline in Cluster of Differentiation 4(CD4) Cell Counts at Week 48 for Both Arms.
Description: The change from baseline in cluster of differentiation 4(CD4) cell counts at week 48 for both arms.
Time Frame: At week 48 of both arms.
Reporting Status: Not Posted

4. Secondary Outcome: The Proportion of Treatment Failure at Week 48 for Both Arms.
Description: The proportion of treatment failure, defined as detectable HIV RNA copies copies/mL, at week 48 for both arms.
Time Frame: At week 48 of both arms
Measure: Count of Participants; unit: Participants
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 51 | 54
Participants | 2 | 2

ADVERSE EVENTS:
Arm/Group | Raltegravir | Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54
Other Adverse Events (participants affected / at risk) | 4/51 | 10/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Raltegravir (N=51) | Efavirenz (N=54)
Insomnia (Nervous system disorders) | 0 | 6
CK Elevation (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Hypertriglycemia (Metabolism and nutrition disorders) | 1 | 0
Swallowing Difficulties (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes